CLINICAL TRIAL: NCT03881501
Title: A Single Arm, Observational Clinical Trial to Evaluate the Efficacy and Safety of Combination Treatment With Sintilimab Injection Plus Endostar in Untreated Locally Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: Evaluate the Treatment With Sintilimab Injection Plus Endostar in Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Head of the cancer center, Huazhong University of Science and Technology
Other Study IDs: TJCC009
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular Carcinoma; Sintilimab Injection; Endostar
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is a a single arm, observational clinical trial to evaluate the efficacy and safety of combination treatment with sintilimab injection plus endostar in untreated locally advanced or metastatic hepatocellular carcinoma.

DETAILED DESCRIPTION:
For the first line treatment with untreated locally advanced or metastatic hepatocellular carcinoma, sintilimab injection plus endostar might be one of the treatment choices.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to comply with the study plans in this protocol and sign the informed consent;
2. Age of 18-75 years;
3. Cytological or histological diagnosis of untreated locally advanced or metastatic hepatocellular carcinoma;
4. Diseases are not suitable for radical surgery and/or local treatment, or disease progression occurs after surgery and/or local treatment;
5. At least one measurable lesion as defined by RECIST 1.1 criteria and untreated lesion;
6. Patients who have received previous local treatment (e.g., radiofrequency ablation, ethanol or acetic acid injection, cryoablation, high intensity focused ultrasound, transcatheter arterial chemoembolization, transcatheter arterial embolization, etc.) are eligible to participate in the study if the target lesion has not received local treatment before, or if the target lesion within the scope of local treatment has subsequently developed on the basis of RECIST v1.1;
7. ECOG performance status of 0-1;
8. Child-Pugh A;
9. Bone marrow function: absolute neutrophil count(ANC) ≥1.5×109 /L, platelet count(PLT) ≥75×109 /L, hemoglobin(HB) ≥90 g/L;
10. alanine glutamate transaminase (ALT) and glutamate transaminase (AST) ≤5 x upper limit of normal range (ULN);total bilirubin (TBIL)≤3 x upper limit of normal range (ULN);Creatinine(Cr)≤1.5 x upper limit of normal range(ULN);Serum albumin (> 28 g/L) (2.8 g/dL);Patients not receiving anticoagulation therapy: INR or aPTT < 2 *ULN;Urinary cellulose test paper results Proteinuria < 2 (7 days before the start of treatment);Patients with baseline cellulose test paper urine test results (> 2 proteinuria) should collect 24-hour urine, and then must confirm that the 24-hour urinary protein content is less than 1 g;
11. HIV test results were negative at screening;
12. Records of virological status of hepatitis, confirmed by serological tests of HBV and HCV;
13. Patients with active hepatitis B virus (HBV) infection:HBV DNA < 500 IU/mL was obtained within 28 days before the start of the study, and received at least 14 days of anti-HBV treatment (based on local standard treatment, such as entecavir) prior to the study, and was willing to continue treatment during the study period.

Exclusion Criteria:

1. Systemic HCC treatment has been received in the past;
2. History of primary immunodeficiency is known;
3. It is known to have active tuberculosis;
4. History of allogeneic organ transplantation and hematopoietic stem cell transplantation is known;
5. It is known that there is a history of human immunodeficiency virus (HIV) infection (that is, HIV antibody positive);
6. Severe allergic/allergic reactions to humanized antibodies or fusion proteins were observed;
7. It is known to have hypersensitivity to any component contained in Endor preparations;
8. Initial serious heart disease patients include congestive heart failure, uncontrollable high-risk arrhythmia, unstable angina pectoris, myocardial infarction, severe valvular disease and refractory hypertension;
9. History of PIA meningitis;
10. Major cardiovascular diseases (e.g. New York Heart Association Grade II or more serious heart disease, myocardial infarction or cerebrovascular accident), unstable arrhythmia or unstable angina pectoris, occurred within three months before the start of treatment;
11. Major surgical treatments (except diagnosis) were received within 4 weeks before the start of the study, or major surgical treatments were expected during the study period;
12. Other malignant tumors were diagnosed within 5 years before the first administration. Exceptions included radical basal cell carcinoma, squamous cell carcinoma, adequately treated cervical cancer in situ, and localized prostate cancer;
13. Active infections requiring systemic treatment;
14. Fiberboard HCC, sarcomatoid HCC or mixed cholangiocarcinoma and HCC are known;
15. Moderate or severe ascites;
16. History of hepatic encephalopathy;
17. Patients with a history of HCV infection but negative results of HCV RNA PCR may consider that they are not infected with HCV;
18. Systemic glucocorticoid therapy or any other form of immunosuppressive therapy is being administered within 7 days prior to the diagnosis of immunodeficiency or the study's first administration; physiological doses of glucocorticoid (<10mg/day prednisone or equivalent) are allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Untreated Locally Advanced or Metastatic Hepatocellular Carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 3 years
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
PFS | up to 3 years
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
OS | up to 3 years
  Overall survival is defined as time from the start of treatment until death due to any reason.
DOR | up to 3 years
  The time between the first recorded and objective remission to the first onset of disease progression or all-cause death (whichever happens first)
Safety as measured by number and grade of adverse events | up to 3 years
  Summary adverse events according to NCI-CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Xianglin Yuan, MD,PhD, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided